CLINICAL TRIAL: NCT07131384
Title: The Interaction Between Inorganic Nitrate Supplementation and Metformin on Exercise Capacity, Vascular Function, and Insulin Sensitivity in Individuals With Pre-Diabetes
Brief Title: Interaction Between Inorganic Nitrate Supplementation and Metformin in Individuals With Prediabetes
Acronym: NO3-PreDM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jason Allen, Professor, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 302659
Record Dates: First submitted 2025-08-06; First posted 2025-08-20 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Males; Females; Sedentary; Metformin; Prediabetes
Keywords: Prediabetic Individuals; Exercise Capacity; Vascular health; Inorganic nitrate; Insulin Sensitivity
MeSH Terms: conditions — Sedentary Behavior; Prediabetic State; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Comparator (Naive to metformin) (Experimental): Participants will supplement with nitrate-rich beetroot juice (BRJ) for 4 days: 6.45 mmol of NO3 in the morning and 6.45 mmol in the evening for 3 days, and 12.9 mmol 2 hours before the lab visit. Supplement order based on randomization and crossover will happen after a minimum of a 7-day washout period.
  Interventions: Dietary Supplement: Dietary Supplement: Inorganic Nitrate (Beetroot juice)
- Placebo Comparator (Naive to metformin) (Placebo Comparator): Participants will supplement with nitrate-depleted beetroot juice (BRJ) for 4 days: 6.45 mmol of NO3 in the morning and 6.45 mmol in the evening for 3 days, and 12.9 mmol 2 hours before the lab visit. Supplement order based on randomization and crossover will happen after a minimum of a 7-day washout period.
  Interventions: Dietary Supplement: Dietary supplement: Placebo (Nitrate-depleted beetroot juice)
- Active Comparator (Taking metformin) (Experimental): Participants will supplement with nitrate-rich beetroot juice (BRJ) for 4 days: 6.45 mmol of NO3 in the morning and 6.45 mmol in the evening for 3 days, and 12.9 mmol 2 hours before the lab visit. Supplement order based on randomization and crossover will happen after a minimum of a 7-day washout period.
  Interventions: Dietary Supplement: Dietary Supplement: Inorganic Nitrate (Beetroot juice)
- Placebo Comparator (Taking metformin) (Placebo Comparator): Participants will supplement with nitrate-depleted beetroot juice (BRJ) for 4 days: 6.45 mmol of NO3 in the morning and 6.45 mmol in the evening for 3 days, and 12.9 mmol 2 hours before the lab visit. Supplement order based on randomization and crossover will happen after a minimum of a 7-day washout period.
  Interventions: Dietary Supplement: Dietary supplement: Placebo (Nitrate-depleted beetroot juice)

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Inorganic Nitrate (Beetroot juice) — Participants will be supplemented with inorganic nitrate in the form of beetroot juice for 4 days (12.9 mmol of NO3/day), and their vascular health, insulin sensitivity, and exercise capacity will be measured post-supplementation. This is a randomized crossover design with 2 parallel groups (Group 1: Currently taking metformin, Group 2: Naive to metformin).
  Arms: Active Comparator (Naive to metformin); Active Comparator (Taking metformin)
Dietary Supplement: Dietary supplement: Placebo (Nitrate-depleted beetroot juice) — Participants will be supplemented with nitrate-depleted beetroot juice for 4 days (<0.01 mmol NO3/day), and their vascular health, insulin sensitivity, and exercise capacity will be measured post-supplementation. This is a randomized crossover design with 2 parallel groups (Group 1: Currently taking metformin, Group 2: Naive to metformin).
  Arms: Placebo Comparator (Naive to metformin); Placebo Comparator (Taking metformin)

SUMMARY:
This study is examining whether short-term supplementation with inorganic nitrate, in the form of beetroot juice, can enhance blood vessel health, insulin sensitivity, and exercise capacity in individuals with prediabetes. We will be comparing the responses in individuals who are taking metformin to those who are naive to metformin. The results from this study may help identify non-pharmacological interventions in prediabetes.

DETAILED DESCRIPTION:
One in 10 Americans have diabetes, with ~ 95% having type 2 diabetes (T2D). Another 1 in 3 have prediabetes, with 70% developing T2D during their lifetimes. Exercise is the standard of care for T2D. However, responses to exercise are blunted in T2D, in part due to the widespread use of metformin, which may inhibit mitochondrial function. Alternative therapies, such as inorganic nitrate supplementation, may provide benefits without attenuating exercise responses.

Purpose: To examine inorganic nitrate supplementation on exercise tolerance, vascular function, and insulin sensitivity in subjects with PD (an ideal time to prevent progression to T2D) who are either taking or naïve to metformin pharmacotherapy.

This study willl recruit twenty-four individuals with PD (12 on, 12 metformin naïve) will participate in a double-blind cross-over design after either oral nitrate or placebo supplementation, including: 1) tests of vascular function (pulse wave velocity, flow mediated dilation, microvascular function with post-occlusive reactive hyperemia, local thermal heating, and skin ACh iontophoresis); 2) exercise testing to determine VO2peak and lactate threshold; 3) an oral glucose tolerance test; and 4) an exercise time trial to exhaustion.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who can communicate meaningfully with the investigator and can provide written consent.
* Confirmed prediabetic individuals (ages 18-60 years old) (2-hour glucose of 140-199 mg/dL following OGTT test or HbA1c between 5.7-6.4% tested on two occasions within 6 months).
* Taking metformin (stable dose for at least a week) or naïve to metformin
* Sedentary (<1 day/week of structured exercise)
* Be able to perform exercise on a cycle ergometer without assistance
* Stable medication regimen for the last 6 months
* If female, have a normal menstrual cycle

Exclusion Criteria:

* Estimated Glomerular filtration rate (GFR) ≤ 45
* Body mass index ≥ 40 Kg/m2
* HbA1c > 6.4%
* Smokers within the last 5 years
* Has experienced significant weight loss ~3 kg in the last three months or is taking any weight loss drugs
* Current medical condition that prohibits exercising at high intensities
* Currently on hormone replacement of any kind
* History of myocardial infarction, cerebrovascular event, acute or unstable disease other than pre-diabetes or obesity
* Currently taking any of the following medications (calcium channel blockers, statins, ACE or renin inhibitors, angiotensin receptor blockers, organic nitrates (e.g., nitroglycerine) or recent regular use of inorganic nitrates, alpha- or beta-blockers, diuretics, proton pump inhibitors, PDE-5 inhibitors (e.g.,: Cialis, Viagra), or xanthine oxidase inhibitors (e.g.,: Allopurinol))
* Oral antibiotic use within the previous four weeks, including over-the-counter antibacterial mouthwash or a mouthwash containing chlorhexidine and unwilling to discontinue use
* Oral cancer/severe oral disease
* Uncontrolled hypertension (>140/90)
* Had hysterectomy or oophorectomy
* Fetuses, neonates, children, prisoners, cognitively impaired, non-English speaking participants

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Vascular Endothelial Function (Pulse wave analysis and velocity [PWA/V]) | 3 days following either active NO3 or placebo without nitrate (following 7-day washout).
  PWA/V- These measures will be calculated using the SphygmoCor XCEL system (AtCor Medical). This system will provide arterial stiffness, central, and peripheral pressure waveforms.
Vascular Endothelial Function (Flow-Mediated Dilation [FMD]) | 3 days following either active NO3 or placebo without nitrate (following 7-day washout).
  FMD- Participants will be placed in a supine position with their left forearm slightly extended and supinated, and their legs straight. The arteries will be imaged using a high-resolution 7.5 MHz linear array transducer at rest, during 5 minutes of forearm occlusion via cuff inflation, and continuously for 3 minutes post-occlusion. An EKG trigger will be used to capture images during the end-diastole of the cardiac cycle.
Skin microvascular function using post-occlusive reactive hyperemia (PORH) | 3 days following either active NO3 or placebo without nitrate (following 7-day washout)
  Skin microvascular function will be measured using Moor Instruments' FLPI-2 laser speckle imaging system. PORH will also be measured during the FMD measurement. Baseline measures will be captured, and the cuff will be inflated for 5 minutes, with the post-occlusion reactive period being measured. The laser positioned above the forearm skin will measure skin blood flow at all these time points.
Skin microvascular function: Change in Skin Microvascular Dilation in Response to Local Thermal Heating | 3 days following either active NO3 or placebo without nitrate (following 7-day washout).
  Skin microvascular function will be measured using Moor Instruments' FLPI-2 laser speckle imaging system. For LTH, ~2 mL of diH2O will be placed on a small disc on the forearm. The solution will be slowly heated to 44 °C. This will allow us to measure the endothelial function of the microcirculation in the skin.
Skin microvascular function: Change in microvascular dilation in response to acetylcholine (ACh) | 3 days following either active NO3 or placebo without nitrate (following 7-day washout)
  Skin microvascular function will be measured using Moor Instruments' FLPI-2 laser speckle imaging system. For skin ACh iontophoresis, ~2 ml of 2% ACh solution (0.1g of ACh in diH2O and filtered) and low current will be used to deliver small quantities of ACh to the skin. This will allow us to measure the endothelial function of the microcirculation in the skin.
Oral Glucose Tolerance Test (OGTT) | 3 days following either active NO3 or placebo without nitrate (following 7-day washout).
  Participants will consume a 75g glucose beverage and then undergo a test to measure insulin, glucose, and C-peptide. A qualified team member will insert a catheter into the antecubital vein for the collection of blood. Blood will be collected at 5 timepoints to estimate insulin sensitivity: before drinking the 75g sugar beverage (0 minutes), and every 30 minutes until the end of the test (120 minutes). Participants will rest in a supine position for the duration of the test.
Plasma Nitrate/Nitrite | 4 days following either active NO3 or placebo without nitrate (following 7-day washout).
  Plasma samples will be collected to assess changes in plasma nitrate and nitrite following either BRJ or placebo.
Cardiorespiratory fitness | 4 days following either active NO3 or placebo without nitrate (following 7 day washout).
  Peak aerobic capacity (VO2peak) will be assessed on a cycle ergometer. An IV will be placed and lactate measured during rest and after the completion of every 3-minute stage to determine VO2 at lactate threshold and VO2peak.
Exercise time trial to exhaustion (TTE) | 4 days following either active NO3 or placebo without nitrate (following 7 day washout).
  Participants will complete a time-to-exhaustion (TTE) test on a cycle ergometer. Participants will begin cycling for 4 minutes at 20 Watts as a warm-up. They will then cycle at a work rate equivalent to 75% of the difference between lactate threshold and VO2peak achieved prior. The TTE test will be terminated when pedal cadence falls ≥ 10 rpm for ≥ 5 sec. When participants reach exhaustion, they will complete a 3-minute unloaded recovery period on the cycle ergometer.
Tissue oxygenation during exercise (near-infrared spectropscopy [NIRS] | 4 days following either active NO3 or placebo without nitrate (following 7-day washout).
  Tissue oxygenation will be captured noninvasively using near-infrared spectrometry (NIRS, PortaMon, Artinis Medical Systems B.V., The Netherlands) positioned on the gastrocnemius (calf) or vastus lateralis (quad) muscle during the VO2peak/lactate test.
Oral nitrate reducing capacity (ONRC) | 4 days following either active NO3 or placebo without nitrate (following 7-day washout).
  To assess the oral microbiome's ability to reduce nitrate to nitrite, the participant will rinse their mouth with a solution of potassium nitrate and ultra-pure water for five minutes. The rinsed solution will be collected into a 50ml Falcon tube. The nitrite concentration will be measured to determine ONRC

SECONDARY OUTCOMES:
Oral Microbiome | 4 days following either active NO3 or placebo without nitrate (following 7-day washout).
  In order to assess abundance and classification of nitrate-reducing bacteria, a sample of the oral microbiome will be obtained. The dorsal surface of the tongue will be swabbed using a 6" HydraFlock Sterile Large Flock Swab for 60 seconds (Puritan Medical Products, USA). Additionally, an unstimulated saliva sample (~5ml) will be collected through an unstimulated drool technique. Both swab and saliva samples will be sequenced to analyze bacteria present in the oral microbiome following supplement/placebo.
Biomarker Analyses: Concentration of Inflammatory markers in fasting blood plasma | Sample collected 4 days post active NO3 juice/placebo and will be analyzed post study completion.
  The investigators plan to assess various markers of inflammation. A fasting blood sample will be collected to measure markers of inflammation.
Biomarker Analyses: Concentration of Oxidative stress markers in fasting blood plasma | Sample collected 4 days post active NO3 juice/placebo and will be analyzed post study completion.
  The investigators plan to assess various markers of oxidative stress. A fasting blood sample will be collected to measure markers of oxidative stress.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Weltman, PhD, Principal Investigator — University of Virginia

IPD SHARING:
Plan to Share IPD: No